CLINICAL TRIAL: NCT05423132
Title: Study on the Efficacy of Infiltration of Upper Cluneal Nerves in Chronic Pain Related to Cluneal Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left the team
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Collaborators: Université Libre de Bruxelles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B0762022220503
Record Dates: First submitted 2022-06-08; First posted 2022-06-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Cluneal Syndrome; Nerve Entrapment Syndrome
Keywords: Superior cluneal nerve entrapment; Chronic Low-back Pain; Injection Site Infiltration; Local anesthetic; Pain; Cluneal nerve block
MeSH Terms: conditions — Charcot-Marie-Tooth Disease; Pain | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiological serum Group (Active Comparator): The cluneal nerve block is performed under ultrasound using the Thomas Dahl Nielsen and Thomas Fichtner Bendtsen method.
  The patients are placed in ventral decubitus. A sensor of high linear frequency is moved toward the middle and posterior to where the aponeurosis of the transverse muscle and the thoraco-lumbar fascia meet, following the appearance of the thoracolumbar fascia and then the appearance of the posterior ilio-costalis muscle under the fascia lumbar area. The infiltration is carried out "in-plane", with a lateral towards the median axis direction, in a way, that it penetrates perpendicularly the fascia
  The physiological serum (NaCl 0.9%) will be injected, on each side, into the aponeurosis and the muscle in the area where the superior cluneal nerves pass. An easy separation of the thoraco- lumbar fascia and the ilio-costalis muscle is achieved during injection by slightly raising the needle towards the median axis as the space opens up gradually.
  Interventions: Drug: Physiological serum injection
- Ropivacaine Group (Experimental): The cluneal nerve block is performed under ultrasound using the Thomas Dahl Nielsen and Thomas Fichtner Bendtsen method.
  The patients are placed in ventral decubitus. A sensor of high linear frequency is moved toward the middle and posterior to where the aponeurosis of the transverse muscle and the thoraco-lumbar fascia meet, following the appearance of the thoracolumbar fascia and then the appearance of the posterior ilio-costalis muscle under the fascia lumbar area. The infiltration is carried out "in-plane", with a lateral towards the median axis direction, in a way, that it penetrates perpendicularly the fascia
  The local anaesthetic (Ropivacaine) will be injected into the aponeurosis and the muscle in the area where the superior cluneal nerves pass. An easy separation of the thoraco- lumbar fascia and the ilio-costalis muscle is achieved during injection by slightly raising the needle towards the median axis as the space opens up gradually.
  Interventions: Drug: Ropivacaine injection

INTERVENTIONS:
Drug: Ropivacaine injection — The patients will receive 15 ml of Ropivacaine 0.375 % on each side.
  Arms: Ropivacaine Group
Drug: Physiological serum injection — The patients will receive 15 ml of physiological serum (NaCl 0.9 %) on each side.
  Arms: Physiological serum Group

SUMMARY:
Lower back pain is a very common complaint in the Chronic Pain Clinic. Its etiology is nonspecific in 85% of the cases. In 1957, Strong and Davila reported that the superior cluneal nerves (SCNs) and middle cluneal nerves (MCNs) can be entrapped around the iliac crest, suggesting a causal relationship between this entrapment (SCN-Entrapment, SCN-E) and low back pain symptom. This is known today as "cluneal syndrome".

Cluneal syndrome remains poorly investigated and is currently a diagnostic challenge. Various types of lumbar movements exacerbate its occurence. The most common theory regarding the origin of this pain evokes that is primarily due to a mechanical cause linked to stenosis or adhesions of fibrous tissue around the cluneal nerves causing distress.

The hypothesis is that the investigator can reduce the pain related to the syndrome of superior cluneal origin thanks to a "volume effect" which aims to detach adhesions and/or aponeurotic stenoses that cause a distress of cluneal nerves.

The aim of this study is to assess the effectiveness of the cluneal nerve block using theThomas Dahl Nielsen ultrasound based technique in patients with chronic low-back pain related to SCN-E. To this end, the investigator will compare physiological serum injection versus local anaesthetic injection, with the aim of reducing short-term pain and improving quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patient signed Inform Consent
2. Patient diagnosed with unilateral or bilateral superior cluneal syndrome :

Diagnostic points will be :

* a maximum pain at the trigger point on the back iliac crest, approximately 7 cm from the median line and 4.5 cm from the poster superior iliac crest. Palpation on this point causes pain reminding the patient's long-term pain),
* Palpation "rolled-palpated" at the buttocks provokes either pain, paraesthesia, or discomfort.
* The criteria of facial syndrome, sacro-iliac syndrome or radiculopathy are excluded.
* Low back pain during back movements.

Exclusion Criteria:

1. Pain not associated to superior cluneal syndrome.
2. Infection at the puncture point.
3. Pain of suspected neoplastic origin.
4. Allergy to local anaesthetics.
5. Refusal of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Reduction of pain intensity in the acute phase of the treatment. | up to 1 hour post-infiltration
  The pain intensity will be assessed using the numeric analogue scale (NAS) at 5 minutes, 30 minutes, 60 minutes and will be compared with (the pain intensity at) the baseline.
  The patient rate the pain from 0 to 10 (0 = no pain; 10 = worst pain imaginable)

SECONDARY OUTCOMES:
Reduction of pain in the late phase of the treatment. | up to 3 months post-infiltration
  The pain intensity will be assessed with the numeric analogue scale (NAS) at 15 days, 1 month, 3 month post-infiltration and will be compared with the pain intensity at the baseline.
  The patient rate the pain from 0 to 10 (0 = no pain; 10 = worst pain imaginable)
Impact of Pain on daily life | up to 3 months post-infiltration
  Impact of pain on daily life will be evaluated according to the Dallas Pain Questionnaire (DPQ).
  The Dallas Pain Questionnaire (DPQ) is 16-item visual analog tool for evaluating how the chronic pain affects the daily activities (The higher the score, the greater the impact of low back pain on quality of life).
  The impact on daily life will be evaluated before infiltration, 15 days, 1 month, 3 months after infiltration.
Incidence of Side effects | up to 3 months post-infiltration
  Side effects will be collected such that the intolerance to the technique and/or injected product, traumatic complications

CONTACTS AND LOCATIONS:
Overall Officials: Panayota Kapessidou, MD,PhD, Study Director — Centre Hospitalier Universitaire Saint Pierre; Walid EL FOUNAS, MD, Principal Investigator — Centre Hospitalier Universitaire Saint Pierre; Aikaterini AMANATIDOU, MD, Principal Investigator — Centre Hospitalier Universitaire Saint Pierre

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Karri J, Singh M, Orhurhu V, Joshi M, Abd-Elsayed A. Pain Syndromes Secondary to Cluneal Nerve Entrapment. Curr Pain Headache Rep. 2020 Aug 21;24(10):61. doi: 10.1007/s11916-020-00891-7. PMID 32821979
- [Background] Randomised trial of ultrasounded guidelines above or cluneal nerve block "Superior Cluneal Nerve Entrapment - Pubmed." Accessed February 7, 2021.
- [Background] Talu GK, Ozyalcin S, Talu U. Superior cluneal nerve entrapment. Reg Anesth Pain Med. 2000 Nov-Dec;25(6):648-50. doi: 10.1053/rapm.2000.18189. PMID 11097676
- [Background] Isu T, Kim K, Morimoto D, Iwamoto N. Superior and Middle Cluneal Nerve Entrapment as a Cause of Low Back Pain. Neurospine. 2018 Mar;15(1):25-32. doi: 10.14245/ns.1836024.012. Epub 2018 Mar 28. PMID 29656623
- [Background] Randomised trial of ultrasound-guided excess cluneal nerve block" Superior Cluneal Nerve Entrapment - Pubmed."
- [Background] Morimoto D, Isu T, Kim K, Imai T, Yamazaki K, Matsumoto R, Isobe M. Surgical treatment of superior cluneal nerve entrapment neuropathy. J Neurosurg Spine. 2013 Jul;19(1):71-5. doi: 10.3171/2013.3.SPINE12420. Epub 2013 Apr 26. PMID 23621641
- [Background] Journal of Prolotherapy "The Management of Cluneal Nerve closed Pain with Prolotherapy," July 10, 2018
- [Background] Hauser RA, Lackner JB, Steilen-Matias D, Harris DK. A Systematic Review of Dextrose Prolotherapy for Chronic Musculoskeletal Pain. Clin Med Insights Arthritis Musculoskelet Disord. 2016 Jul 7;9:139-59. doi: 10.4137/CMAMD.S39160. eCollection 2016. PMID 27429562